CLINICAL TRIAL: NCT01739673
Title: Ultraviolet-A and Riboflavin Treatment for Infectious Keratitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cxlusa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iCXL
Record Dates: First submitted 2012-11-27; First posted 2012-12-03 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2015-08

CONDITIONS: Infectious Keratitis
Keywords: Infectious Keratitis
MeSH Terms: interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultraviolet-A and riboflavin (Experimental)
  Interventions: Other: Ultraviolet-A and riboflavin

INTERVENTIONS:
Other: Ultraviolet-A and riboflavin

SUMMARY:
This study is to evaluate the efficacy of ultraviolet-A (UVA) and riboflavin application (also often referred to as corneal collagen crosslinking) as a method to enhance treatment of infectious keratitis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Ability to provide written informed consent.
3. Likely to complete all study visits.
4. Subjects must have one eye that with a diagnosis of infectious keratitis.

Exclusion Criteria:

1. A corneal perforation.
2. Descemetocele.
3. Pregnancy or breastfeeding.
4. Active Herpes corneal disease.
5. Patient is unwilling or unable to comply with a medication regimen and follow up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Resolution of Signs and Symptoms of Infectious Keratitis | Subjects will be followed until resolution of signs and symptoms, an expected average of 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Study Director — Center For Excellence In Eye Care
Locations (6):
- United States (6):
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Davidorf Eye Group, West Hills, California
  - Corneal Consultants of Colorado, PC, Littleton, Colorado
  - Center for Excellence in Eye Care, Miami, Florida
  - Minnesota Eye Consultants, Minneapolis, Minnesota
  - Ophthalmology Associates, St Louis, Missouri